CLINICAL TRIAL: NCT00174213
Title: Validity and Reliability in Measuring Iliotibial Tract by Using Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701066
Record Dates: First submitted 2005-09-14; First posted 2005-09-15 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 1994-08

CONDITIONS: Knee Injuries
Keywords: iliotibial tract
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to estimate the validity and reliability in measuring the iliotibial tract by using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee injuries who need magnetic resonance imaging (MRI) evaluation

Exclusion Criteria:

* Patients who have an iliotibial tract lesion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1994-09

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Kuo Wang, PhD, Study Director — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, NTU, Taiwan, Taipei, Taiwan